CLINICAL TRIAL: NCT03444675
Title: A Multi-centre, Longitudinal (Cohort) Study in Patients Undergoing Intestinal or Multivisceral Transplantation to Validate Gothenburg Intestinal Transplant Endoscopy Score (GITES) and Evaluate Its Clinical Performance
Brief Title: The Endoscopic Assesment of Intestinal Grafts
Acronym: INTEGRATE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sahlgrenska University Hospital (Other)
Collaborators: Favaloro Foundation University Hospital, Buenos Aires, Argentina (Unknown); MedStar Georgetown University Hospital, Washington DC (Unknown); Hospital Universitario La Paz (Other)
Responsible Party: Principal Investigator, Mihai Oltean, Dr., Sahlgrenska University Hospital
Other Study IDs: GBG18001
Record Dates: First submitted 2018-02-19; First posted 2018-02-23 (Actual); Last update posted 2020-05-15 (Actual); Status verified 2020-05

CONDITIONS: Transplant; Intestine; Transplant; Complication, Rejection; Transplant; Failure, Bowel; Enteritis; Mucosal Inflammation
Keywords: Transplantation; intestine; endoscopy; severity score; transplant rejection; transplant; complications
MeSH Terms: conditions — Rejection, Psychology; Enteritis; Mucositis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study validates prospectively a new endoscopic scoring system (Gothenburg Intestinal Transplant Endoscopy Score, GITES) designed to summarize and stratify the abnormal ileal endoscopic findings after intestinal transplantation. GITES is a five-tier, four grade score which asseses mucosal friability, mucosal erythema and mucosal injury (ulcerations) as well as villous changes according to severity. These features (i.e., endoscopic descriptors) are also grouped from mild to very severe in the same sequence as observed during the progression of several pathologic conditions encountered after intestinal transplantation (acute rejection, infectious enteritis).

ELIGIBILITY:
Inclusion Criteria:

* transplantation of a segment of small intestine (as isolated graft or together with other organs)

Exclusion Criteria:

* contraindications for ileoscopy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients (pediatric or adult) undergoing intestinal transplantation (isolated intestine, liver-intestine, multivisceral, including colon or other organs) irrespective of diagnosis; patients already transplanted can also be included.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2014-04-29 (Actual); Primary Completion 2022-05-01 (Estimated); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
Endoscopic evaluation | 7 years
  To validate the GITES grading system in intestinal graft recipients using high-definition white light endoscopy

SECONDARY OUTCOMES:
Correlations with histology and Clinical course | 1 year
  Comparison and correlation of clinical and histopathological data with endoscopic findings to evaluate the conditions leading to the mucosal alterations defined by established endoscopic descriptors and GITES.
Performance of the grading score | 1 year
  Endpoints include sensitivity, specificity, positive predictive value, negative predictive value as well as inter- and intraobserver variation in the evaluation of the mucosal alterations by means of GITES and using high-definition white light endoscopy;

CONTACTS AND LOCATIONS:
Locations (4):
- MedStar Georgetown University Hospital, Washington D.C., District of Columbia, United States
- Favaloro Foundation University Hospital, Buenos Aires, Argentina
- Hospital Universitario "La Paz", Madrid, Spain
- Sahlgrenska University Hospital, Gothenburg, Sweden

REFERENCES:
- [Background] Sigurdsson L, Reyes J, Putnam PE, del Rosario JF, Di Lorenzo C, Orenstein SR, Todo S, Kocoshis SA. Endoscopies in pediatric small intestinal transplant recipients: five years experience. Am J Gastroenterol. 1998 Feb;93(2):207-11. doi: 10.1111/j.1572-0241.1998.00207.x. PMID 9468243
- [Background] Tabasco-Minguillan J, Weber K, Nelson F, Hutson W, Furukawa H, Abu-Elmagd K, Todo S, Rakela J. Variability in the interpretations of endoscopic findings in patients with intestinal transplantation. Transplant Proc. 1996 Oct;28(5):2775-6. No abstract available. PMID 8908053
- [Background] Varkey J, Stotzer PO, Simren M, Herlenius G, Oltean M. The endoscopic surveillance of the transplanted small intestine: a single center experience and a proposal for a grading score. Scand J Gastroenterol. 2018 Feb;53(2):134-139. doi: 10.1080/00365521.2017.1411523. Epub 2017 Dec 12. PMID 29233031